CLINICAL TRIAL: NCT01551498
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Trial to Evaluate the Safety and Potential Effects of the Dietary Supplement Anatabloc on Antithyroid Autoantibodies and Thyroid Function in Autoimmune Thyroiditis
Brief Title: Evaluating the Dietary Supplement Anatabloc in Thyroid Health-ASAP (Antabloc Supplementation Autoimmune Prevention)
Acronym: ASAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rock Creek Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCP-007
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Thyroiditis, Autoimmune
Keywords: Hashimoto Disease; Thyroiditis
MeSH Terms: conditions — Thyroiditis, Autoimmune; Hashimoto Disease; Thyroiditis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): subject takes one oral placebo lozenge, three times per day
  Interventions: Dietary Supplement: Placebo
- Anatabloc Supplement (Active Comparator): subject takes one oral Supplement lozenge, three time per day
  Interventions: Dietary Supplement: Anatabloc Supplement

INTERVENTIONS:
Dietary Supplement: Anatabloc Supplement — Product, as mint-flavored lozenges (3 mg anatabine per lozenge), to be taken 3 times each day
  Arms: Anatabloc Supplement
Dietary Supplement: Placebo — Placebo, as mint flavored lozenges, to be taken 3 times each day
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety, tolerability, and potential effects of Anatabloc dietary supplementation on antithyroid autoantibodies, thyroid structure, and thyroid function in subjects with autoimmune thyroiditis.

DETAILED DESCRIPTION:
This is a 5-visit, 12-week, double-blind, randomized, placebo-controlled, parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-70 years of age
* having positive antibodies against thyroid peroxidase
* having sonographic evidence consistent with a diagnosis of Hashimoto's thyroiditis

Exclusion Criteria:

* having evidence of end-stage thyroiditis
* being a current smoker or smokeless tobacco user
* be taking systemic glucocorticoids, interferon-alpha, anti-CD20 antibody, or anti-CTLA-4 antibody
* be taking any medication for treatment of autoimmune thyroiditis other than L-thyroxine or equivalent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Numbers of subjects experiencing adverse effects as a measure of safety | 3 months
  Collected data on the numbers and types of any adverse effects related to the use of Anatabloc by subjects

SECONDARY OUTCOMES:
Measured changes in markers of autoimmune thyroiditis: changes in blood levels of anti-thyroid auto-antibodies, and changes in the volume and vascularization of the thyroid | 3 months
  To determine if dietary supplementation with Anatabloc has an effect on antithyroid autoantibody levels, thyroid structure, and/or thyroid function in subjects with autoimmune thyroiditis

CONTACTS AND LOCATIONS:
Overall Officials: Maria Varga, MD, Study Director — Star Scientific, Inc
Locations (9):
- United States (9):
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Robert J. Becker, M.D., LTD, La Grange, Illinois
  - Associated Endocrinologists, P.C., West Bloomfield, Michigan
  - New Jersey Physicians, LLC, Clifton, New Jersey
  - Texas Diabetes & Endocrinology, Austin, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas

REFERENCES:
- [Derived] Schmeltz LR, Blevins TC, Aronoff SL, Ozer K, Leffert JD, Goldberg MA, Horowitz BS, Bertenshaw RH, Troya P, Cohen AE, Lanier RK, Wright C 4th. Anatabine supplementation decreases thyroglobulin antibodies in patients with chronic lymphocytic autoimmune (Hashimoto's) thyroiditis: a randomized controlled clinical trial. J Clin Endocrinol Metab. 2014 Jan;99(1):E137-42. doi: 10.1210/jc.2013-2951. Epub 2013 Dec 20. PMID 24178792